CLINICAL TRIAL: NCT07251088
Title: Dyadic, App-supported Collaborative Care Intervention Trial for Family Caregivers of People Living With Dementia - The Multi-center Living@Home Study
Brief Title: Dyadic, App-supported Collaborative Care Intervention Trial for Family Caregivers of People Living With Dementia
Acronym: Living@Home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University Medicine Rostock, Rostock (Unknown); AGAPLESION ELISABETHENSTIFT gGmbH (Unknown); AOK - Die Gesundheitskasse für Niedersachsen (Unknown); Gemeinnützige Gesellschaft für Psychiatrie Reutlingen mbH (Unknown); Georg-August-Universität Göttingen (Unknown); IKK gesund plus (Unknown); Karlsruher Institut für Technologie (Unknown); Otto-von-Guericke-Universität Magdeburg (Unknown); Universität Konstanz (Unknown); Universität zu Köln (Unknown); University Medicine Greifswald (Other); Federal Joint Committee (Other Government)
Responsible Party: Principal Investigator, Bernhard Michalowsky, Research Group leader, German Center for Neurodegenerative Diseases (DZNE)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01NVF24315
Record Dates: First submitted 2025-09-30; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Dementia; Nurse Care Coordination; Informal Caregiver
Keywords: Dementia; Dementia Care; Caregiver of people with dementia; Dyade; digital health intervention
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Specially qualified nurses (caregiver experts) will provide individualized dementia care management to dyads in the intervention group over a period of twelve months, with the aim of identifying and effectively addressing the unmet needs of both people living with dementia (PlwD) and their caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention): Care as usual
- Individualized Dementia Care Management (Experimental): Dyads in the intervention group will receive individualized dementia care management over a twelve-month period, with the objective of identifying and effectively addressing the unmet needs of people living with dementia (PlwD) and their caregivers. The intervention is complemented by a mobile health application used by both caregivers and Care Specialists, providing caregivers with continuous access to care managers and memory clinics whenever challenges or burdens arise. The app facilitates ongoing monitoring of caregivers' health status and burden through regular realtime data collection, aggregation, and transmission to the care manager, thereby enabling timely and needs-based interventions or re-interventions. Consequently, the frequency and intensity of the intervention are tailored to the dyads' individual circumstances and reported levels of burden.
  Interventions: Other: Experimental arm

INTERVENTIONS:
Other: Experimental arm — Dyads in the intervention group will receive individualized dementia care management over a twelve-month period, with the objective of identifying and effectively addressing the unmet needs of people living with dementia (PlwD) and their caregivers. The intervention is complemented by a mobile health application used by both caregivers and Care Specialists, providing caregivers with continuous access to care managers and memory clinics whenever challenges or burdens arise. The app facilitates ongoing monitoring of caregivers' health status and burden through regular real-time data collection, aggregation, and transmission to the care manager, thereby enabling timely and needs-based interventions or re-interventions. Consequently, the frequency and intensity of the intervention are tailored to the dyads' individual circumstances and reported levels of burden.
  Other Names: Individualized Dementia Care Management
  Arms: Individualized Dementia Care Management

SUMMARY:
In Germany, approximately 1.8 million individuals are living with dementia, representing a considerable share of those requiring long-term care. Many people with dementia (PlwD) express the desire to remain in their home environment for as long as possible. However, the progressive cognitive and physical decline associated with the disease renders caregiving increasingly time-intensive and places a substantial burden on family members. In the absence of sufficient support structures, maintaining home-based care becomes difficult, creating additional strain on the health care system.

The study aims to address these challenges through an innovative intervention. Its primary objectives are: (1) to evaluate whether a dyadic care management model, delivered by specialized nurses with expertise in dementia care and supported by a mobile health application that provides direct access to caregiving experts and memory clinics, can help stabilize the home care situation; (2) to determine whether this approach reduces caregiver burden; and (3) to assess its effectiveness in alleviating neuropsychiatric symptoms in PlwD, compared to usual care.

DETAILED DESCRIPTION:
In Germany, approximately 84% of the five million individuals in need of care are supported at home by informal caregivers, most commonly family members. Only 21% receive professional assistance from care or support services, highlighting the substantial responsibility placed on families. People living with dementia (PlwD) constitute a particularly large share of these care recipients. On average, they require around 36 hours of informal care per week-considerably more than individuals affected by conditions such as cancer (16 hours/week) or stroke (24 hours/week).

Both PlwD and their caregivers, often conceptualized as a dyad, frequently express a strong preference for remaining in their home environment and sustaining home-based care for as long as possible. While many caregivers provide support over extended periods and may even perceive their role as meaningful, the progressive cognitive and physical decline of PlwD, combined with neuropsychiatric symptoms and caregivers' perceived sense of obligation, can result in considerable psychological and physical strain. Such strain is commonly associated with depression, anxiety, diminished subjective well-being, reduced self-efficacy, and social withdrawal. Consequently, the sustainability of home care is often precarious. Indeed, 40% of caregivers of community-dwelling PlwD report being unable to maintain care for longer than one year, leading to institutionalization.

Although support services for caregivers have been steadily expanded in recent years, their utilization remains limited. Barriers include a lack of awareness, organizational hurdles, and, paradoxically, the high demands of caregiving itself, which can hinder access to such services. In the absence of sufficient support, informal care is increasingly substituted by professional long-term care, thereby intensifying pressure on already limited workforce and financial resources within the health care system. This transition is also frequently accompanied by feelings of guilt among caregivers.

Evidence regarding the effectiveness of interventions to support caregivers is mixed. Randomized controlled trials have only partly demonstrated significant reductions in caregiver burden. A meta-analysis indicated that individualized, structured multicomponent interventions-comprising various support modules-are most effective. While there is some evidence for cost-effectiveness, it is constrained by small sample sizes. A model-based analysis suggests that dyadic interventions, which target both PlwD and caregivers, may prolong the feasibility of home-based care and could be cost-effective. However, findings remain inconsistent: a meta-analysis of randomized controlled trials reported positive outcomes in 13 studies but no effect in 9 others. Effectiveness appears to depend strongly on the duration and intensity of interventions. One explanation may be that caregiver needs during periods of heightened burden were not adequately or promptly addressed.

Digital health interventions, such as remote, app-based solutions, offer the potential to overcome these limitations by providing flexible and immediate support at critical moments. Nevertheless, research in this field remains limited, and it is still unclear to what extent digital approaches can stabilize home care situations for PlwD and their families.

ELIGIBILITY:
Inclusion Criteria:

* formal dementia diagnosis
* living in their own home for the person with dementia
* access to a smartphone and internet for the informal caregiver
* informed consent of the participant

Exclusion Criteria:

* not able to provide written consent
* if a legal representative is present, they may give their consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Stability of the home care arrangement (Perseverance Time Scale) | 12 months after baseline assessment
  For the Perseverance Time Scale, informal caregivers are asked (self-assessment) to estimate how long they believe they can continue to provide informal care and, thus, their current care situation. Response options are: less than one week, less than one month, less than six months, less than one year, less than two years, and two years or more.
  This measure is central to evaluating the long-term stability of home-based care - an essential aspect of dementia care, given the chronic and progressive nature of the disease.
Neuropsychiatric symptoms (NPI-Q) | 12 months after baseline assessment
  Another primary outcome is the presence of neuropsychiatric symptoms in PlwD, assessed with the Neuropsychiatric Inventory Questionnaire (NPI-Q), completed by the informal caregiver via face-to-face interviews with the study nurse. Neuropsychiatric symptoms are well-documented contributors to caregiver burden, underlining the dyadic nature of selected primary outcomes. Each of the 12 domains of the NPI-Q includes a survey item that captures the key symptom associated with that domain. For each question, respondents indicate whether the symptom has been present ("Yes") or absent ("No"). If the response is "No," the informant proceeds to the next item. If "Yes," they are asked to rate the severity of the symptom experienced during the past month on a 3-point scale, as well as the caregiver distress caused by the symptom on a 5-point scale. The NPI score can becalculated by adding the scores of the first 10 ir 12 items, higher scores indicate higher presence of psychopathology.
Caregiver burden (ZBI) | 12 months after baseline assessment
  The third primary outcome is the caregiver burden itself, measured via the Zarit Burden Interview (12-item version), which will be self-completed by caregivers. This tool is among the most commonly applied instruments in informal dementia caregiver research, enabling comparability across studies. While the most commonly used form of the Zarit Burden Interview is a 22-item version, the shortened 12-item version has demonstrated comparable psychometric properties (Bedard et al., 2001), offering a time-efficient alternative that reduces respondent burden. Each item on the interview is a statement which the caregiver is asked to rate using a 5-point scale. Response options range from 0 (never) to 4 (nearly always). The result of the instrument is a sum between 0 and 48, higher results indicate a higher subjective level of burden.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Michalowsky, PD Dr. Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (12):
- Germany (12):
  - Institut für Technik der Informationsverarbeitung, Karlsruhe, Baden-Wurttemberg
  - Universität Konstanz, Konstanz, Baden-Wurttemberg
  - Gemeinnützige Gesellschaft für Psychiatrie Reutlingen mbh, Reutlingen, Baden-Wurttemberg
  - AGAPLESION Elisabethenstift, Darmstadt, Hesse
  - AOK Niedersachsen, Hanover, Lower Sachsony
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - DZNE, Greifswald, Mecklenburg-Vorpommern
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Universität zu Köln, Cologne, North Rhine-Westphalia
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg, Saxony
  - IKK gesund plus, Magdeburg, Saxony

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scharf A, Michalowsky B, Radke A, Kleinke F, Schade S, Platen M, Buchholz M, Pfaff M, Iskandar A, van den Berg N, Hoffmann W. Identifying and Addressing Unmet Needs in Dementia: The Role of Care Access and Psychosocial Support. Int J Geriatr Psychiatry. 2025 Apr;40(4):e70066. doi: 10.1002/gps.70066. PMID 40148225
- [Background] Eichler T, Thyrian JR, Hertel J, Richter S, Wucherer D, Michalowsky B, Teipel S, Kilimann I, Dreier A, Hoffmann W. Unmet Needs of Community-Dwelling Primary Care Patients with Dementia in Germany: Prevalence and Correlates. J Alzheimers Dis. 2016;51(3):847-55. doi: 10.3233/JAD-150935. PMID 26890767
- [Background] Michalowsky B, Eichler T, Thyrian JR, Hertel J, Wucherer D, Laufs S, Flessa S, Hoffmann W. Medication cost of persons with dementia in primary care in Germany. J Alzheimers Dis. 2014;42(3):949-58. doi: 10.3233/JAD-140804. PMID 25125471
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Scharf A, Kleinke F, Michalowsky B, Radke A, Pfitzner S, Muhlichen F, Buchholz M, van den Berg N, Hoffmann W. Sociodemographic and Clinical Characteristics of People Living with Dementia and Their Associations with Unmet Healthcare Needs: Insights from the Baseline Assessment of the InDePendent Study. J Alzheimers Dis. 2024;99(2):559-575. doi: 10.3233/JAD-231173. PMID 38669533
- [Background] Kleinke F, Michalowsky B, Radke A, Platen M, Muhlichen F, Scharf A, Mohr W, Penndorf P, Bahls T, van den Berg N, Hoffmann W. Advanced nursing practice and interprofessional dementia care (InDePendent): study protocol for a multi-center, cluster-randomized, controlled, interventional trial. Trials. 2022 Apr 11;23(1):290. doi: 10.1186/s13063-022-06249-1. PMID 35410437